CLINICAL TRIAL: NCT02419157
Title: Effectiveness of One- and Two-step Self-etching Adhesives Applied With or Without Selective Enamel Etching: a 2-year Randomized Controlled Clinical Trial
Brief Title: Selective Enamel Etching in Self-etching Adhesives: a 2-year Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Caroline Ely, Associate Faculty, University of Guarulhos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRGRE 2015
Record Dates: First submitted 2015-03-29; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Selective Enamel Etching in Dental Restorations
Keywords: Cervical lesions; Clinical trial; Self-etch adhesive
MeSH Terms: interventions — phosphoric acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clearfil SE Bond Etch (CSE-E) (Active Comparator): CSE-E (n=28): After shade selection, teeth were restored under relative isolation. Lesions were cleaned with pumice and water in a rubber cup followed by rinsing and drying. An enamel bevel of 1-2 mm was prepared with a diamond bur operated in a high-speed handpiece under air-water spray. Enamel margins were selectively etched with 36% phosphoric acid for 15s and subsequently thoroughly rinsed and air-dried. Adhesive system was applied according to manufacturers' instructions and light-cured with an LED for 10s. NCCLs were restored incrementally with a microhybrid composite resin. Increments were light cured for 20s. Afterwards, retraction cord was removed and finishing and polishing were performed with rubber points.
  Selective enamel etching with 36% phosphoric acid
  Interventions: Drug: Selective enamel etching with 36% phosphoric acid; Device: Clearfil SE Bond
- Xeno V+ Etch (XV-E) (Active Comparator): XV-E (n=28): After shade selection, teeth were restored under relative isolation. Lesions were cleaned with pumice and water in a rubber cup followed by rinsing and drying. An enamel bevel of 1-2 mm was prepared with a diamond bur operated in a high-speed handpiece under air-water spray. Enamel margins were selectively etched with 36% phosphoric acid for 15s and subsequently thoroughly rinsed and air-dried. Adhesive system was applied according to manufacturers' instructions and light-cured with an LED for 10s. NCCLs were restored incrementally with a microhybrid composite resin. Increments were light cured for 20s. Afterwards, retraction cord was removed and finishing and polishing were performed with rubber points.
  Selective enamel etching with 36% phosphoric acid
  Interventions: Drug: Selective enamel etching with 36% phosphoric acid; Device: Xeno V
- Clearfil SE Bon Non-etch (CSE-NE) (Active Comparator): CSE-NE (n=28): After shade selection, teeth were restored under relative isolation. Lesions were cleaned with pumice and water in a rubber cup followed by rinsing and drying. An enamel bevel of 1-2 mm was prepared with a diamond bur operated in a high-speed handpiece under air-water spray. Adhesive system was applied according to manufacturers' instructions and light-cured with an LED for 10s. NCCLs were restored incrementally with a microhybrid composite resin. Increments were light cured for 20s. Afterwards, retraction cord was removed and finishing and polishing were performed with rubber points.
  No selective enamel etching with 36% phosphoric acid
  Interventions: Drug: No selective enamel etching with 36% phosphoric acid; Device: Clearfil SE Bond
- Xeno V+ Non-etch (XV-NE) (Active Comparator): XV-NE (n=28): After shade selection, teeth were restored under relative isolation. Lesions were cleaned with pumice and water in a rubber cup followed by rinsing and drying. An enamel bevel of 1-2 mm was prepared with a diamond bur operated in a high-speed handpiece under air-water spray. Adhesive system was applied according to manufacturers' instructions and light-cured with an LED for 10s. NCCLs were restored incrementally with a microhybrid composite resin. Increments were light cured for 20s. Afterwards, retraction cord was removed and finishing and polishing were performed with rubber points.
  No selective enamel etching with 36% phosphoric acid
  Interventions: Drug: No selective enamel etching with 36% phosphoric acid; Device: Xeno V

INTERVENTIONS:
Drug: Selective enamel etching with 36% phosphoric acid — Etch: selective 36% phosphoric acid enamel etching
  Other Names: 36% phosphoric acid
  Arms: Clearfil SE Bond Etch (CSE-E); Xeno V+ Etch (XV-E)
Drug: No selective enamel etching with 36% phosphoric acid — Non-etch: without phosphoric acid selective enamel etching
  Other Names: Without 36% phosphoric acid
  Arms: Clearfil SE Bon Non-etch (CSE-NE); Xeno V+ Non-etch (XV-NE)
Device: Clearfil SE Bond
  Arms: Clearfil SE Bon Non-etch (CSE-NE); Clearfil SE Bond Etch (CSE-E)
Device: Xeno V
  Arms: Xeno V+ Etch (XV-E); Xeno V+ Non-etch (XV-NE)

SUMMARY:
The purpose of this study is to evaluate the clinical effectiveness of non-carious cervical lesions (NCCLs) restored with two self-etching adhesive systems applied with or without selective enamel etching.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical effectiveness of non-carious cervical lesions (NCCLs) restored with two self-etching adhesive systems: Clearfil SE Bond (Kuraray Noritake, Japan) and Xeno V + (Dentsply De Trey, Germany) applied with or without 36% phosphoric acid enamel etching. Assessments were at baseline, 3, 6, 12, 18 and 24 months of clinical service.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years;
* Present at least 4 NCCLs in vital teeth with margins in enamel and dentin (and its largest area in dentin), independently of teeth location;
* Non-smoking;
* Read and sign the Statement of Informed Consent.

Exclusion Criteria:

* Compromised medical history;
* Severe or chronic periodontitis;
* Extreme caries sensitivity;
* Heavy bruxism;
* Under orthodontic treatment;
* Poor oral hygiene;
* Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Restoration retention rate as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Restoration marginal integrity as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months
Restoration marginal staining as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months
Secondary caries as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months
Post-operative sensitivity as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months
Pulp vitality as measured by modified U.S. Public Health Service evaluation criteria at baseline, 3, 6, 12, 18 and 24 months | Baseline, 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: André F Reis, Principal Investigator — University of Guarulhos

REFERENCES:
- [Background] De Munck J, Van Landuyt K, Peumans M, Poitevin A, Lambrechts P, Braem M, Van Meerbeek B. A critical review of the durability of adhesion to tooth tissue: methods and results. J Dent Res. 2005 Feb;84(2):118-32. doi: 10.1177/154405910508400204. PMID 15668328
- [Background] De Munck J, Vargas M, Iracki J, Van Landuyt K, Poitevin A, Lambrechts P, Van Meerbeek B. One-day bonding effectiveness of new self-etch adhesives to bur-cut enamel and dentin. Oper Dent. 2005 Jan-Feb;30(1):39-49. PMID 15765956
- [Background] Perdigao J, Geraldeli S. Bonding characteristics of self-etching adhesives to intact versus prepared enamel. J Esthet Restor Dent. 2003;15(1):32-41; discussion 42. doi: 10.1111/j.1708-8240.2003.tb00280.x. PMID 12638771
- [Background] Peumans M, De Munck J, Van Landuyt K, Lambrechts P, Van Meerbeek B. Five-year clinical effectiveness of a two-step self-etching adhesive. J Adhes Dent. 2007 Feb;9(1):7-10. PMID 17432395
- [Background] Van Meerbeek B, Kanumilli P, De Munck J, Van Landuyt K, Lambrechts P, Peumans M. A randomized controlled study evaluating the effectiveness of a two-step self-etch adhesive with and without selective phosphoric-acid etching of enamel. Dent Mater. 2005 Apr;21(4):375-83. doi: 10.1016/j.dental.2004.05.008. PMID 15766585
- [Background] Reis AF, Bedran-Russo AK, Giannini M, Pereira PN. Interfacial ultramorphology of single-step adhesives: nanoleakage as a function of time. J Oral Rehabil. 2007 Mar;34(3):213-21. doi: 10.1111/j.1365-2842.2006.01656.x. PMID 17302950
- [Background] Cvar JF, Ryge G. Reprint of criteria for the clinical evaluation of dental restorative materials. 1971. Clin Oral Investig. 2005 Dec;9(4):215-32. doi: 10.1007/s00784-005-0018-z. No abstract available. PMID 16315023